CLINICAL TRIAL: NCT02931474
Title: The Impact of GHRH on Sleep Promotion and Endocrine Regulation in Service Members Who Sustained a Traumatic Brain Injury and Have Current Insomnia
Brief Title: Impact of GHRH on Sleep Promotion and Endocrine Regulation in Service Members Who Sustained a Traumatic Brain Injury and Have Current Insomnia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 170005; 17-NR-0005
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2017-03-08

CONDITIONS: Sleep Disorder; Traumatic Brain Injury
Keywords: Growth Hormone; Traumatic Brain Injury; Insomnia; Polysomnography; NREM Sleep
MeSH Terms: conditions — Sleep Wake Disorders; Brain Injuries, Traumatic; Sleep Initiation and Maintenance Disorders | interventions — tesamorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Salt Water Solution
  Interventions: Other: Placebo
- Tesamorelin (Experimental): Growth Hormone-Releasing
  Interventions: Drug: Tesamorelin

INTERVENTIONS:
Drug: Tesamorelin — Growth Hormone-Releasing
  Arms: Tesamorelin
Other: Placebo
  Arms: Placebo

SUMMARY:
Background:

People who have had a traumatic brain injury (TBI) often have trouble sleeping. TBI may also alter hormones, which can cause poor sleep. Researchers believe that a form of growth hormone releasing hormone (GHRH) might improve sleep in service members and veterans who have had a TBI.

Objective:

To see if GHRH can improve sleep in people who have had a TBI.

Eligibility:

Active duty service members or veterans (active duty in the past 10 years) ages 18-45 who have had a TBI in the past 6 months to 10 years.

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Getting ACTH (a hormone) through an intravenous catheter (thin plastic tube)

Interview about their mood and alcohol and drug use

Questionnaires about their TBI, mood, and sleep

Participants will have 2 overnight study visits a couple weeks apart. These will include:

Physical exam

Urine sample

Two intravenous catheters placed. Blood samples will be taken throughout the night.

Two shots under the skin of the belly. The shots will be GHRH on one visit and placebo on the other.

Spending the night in the sleep lab. Their brain waves will be recorded with electrodes placed on the scalp.

A questionnaire in the morning about their sleep

Participants will be called a few days after each overnight visit. They will be asked about how they are feeling and to rate their sleep.

DETAILED DESCRIPTION:
Objective: Traumatic brain injury (TBI) is the hallmark injury of deployment in Iraq and Afghanistan. Up to one-third of service members who sustain a TBI are diagnosed with a sleep disorder; insomnia being one of the most common. Currently, over half of TBI-associated insomnia cases remain untreated due to poor efficacy of available pharmacologic agents. Neuroendocrine dysfunction is an important mechanism linking TBI and disordered sleep, thus pharmacological agents that address this dysfunction may be effective in treating TBI-related insomnia. The neuroendocrine system is essential for regulating sleep and circadian function. Decreased neuroendocrine function, including the hypothalamus and the somatotrophic cells of the anterior pituitary, which regulate growth hormone secretion, likely contributes to insomnia. This assertion is supported by previous studies that demonstrated the sleep-promoting effects of growth hormone releasing hormone (GHRH) administration in healthy controls, the elderly, and participants with depression. Therefore, we propose that administration of GHRH will address the underlying mechanisms of insomnia in service members and veterans who sustained a TBI, and provide a pharmacological agent more robust than currently available treatments.

Study population: This study will recruit 50 active duty service members and veterans with a documented TBI to participate in one of two study groups. The insomnia group (n=25) will include participants that have a current clinical diagnosis of insomnia without obstructive sleep apnea. The no-insomnia group (n=25) will include participants with no current clinical diagnosis of insomnia or obstructive sleep apnea. Withdrawals/dropouts will be replaced to obtain 20 participants per group who complete the study.

Design: A double-blind, randomized, crossover design will be used to examine the impact of tesamorelin (GHRH (1-44) analog) or placebo on total non-rapid eye movement (NREM) time evaluated during two polysomnography visits, scheduled 1-3 weeks apart. Serial blood draws will be obtained during the polysomnography to examine endocrine function and neuropeptide release.

Outcome measures: The primary outcome is change in NREM time following tesamorelin administration compared to placebo. The secondary outcomes are (1) within and between group differences in plasma concentration levels of neuroendocrine proteins following tesamorelin administration compared to placebo and (2) within and between group differences in urinary concentration levels of growth hormone following tesamorelin administration compared to placebo.

ELIGIBILITY:
* INCLUSION CRITERIA:

Both groups may be eligible for this research study if they:

1. Are between 18 and 45 years of age (on Visit 1)
2. Are active duty service members or veterans who were active duty within the past 10 years (on Visit 1)
3. Are able to provide medical records documenting a TBI, which occurred within the past 6 months to 10 years (on Visit 1)
4. Are able to provide their own consent
5. Are able to understand the study, as shown by scoring a 6 out of 6 on a consent quiz
6. (For women only) agree not to breastfeed from the time of enrollment in the study until 1 month after the last exposure to tesamorelin
7. (For women of childbearing potential only) have a negative urine pregnancy test and agree to use two effective methods of contraception from the time of enrollment in the study until 1 month after the last exposure to tesamorelin

The insomnia group may be eligible for this research study if they:

1. Have a current clinical diagnosis of insomnia determined by polysomnography
2. Have a PSQI score greater than 10

The no-insomnia group may be eligible for this research study if they:

1. Have no current clinical diagnosis of insomnia determined by self-report
2. Have a PSQI score less than or equal to 5

EXCLUSION CRITERIA:

Both groups may not be eligible for this research study if they:

1. Have obstructive sleep apnea determined by polysomnography (insomnia group) or selfreport (no-insomnia group)
2. Have a known hypersensitivity to tesamorelin and/or mannitol
3. Have taken any of the following medications within the past 30 days: benzodiazepines (e.g., Valium, Ativan, etc.); benzodiazepine receptor agonists (e.g., Ambien, Lunesta, etc.); opiates (e.g., Codeine, Percocet, etc.); or sedatives (e.g., Amytal, Numbutal, etc.)
4. Cannot abstain from using stimulants such as amphetamines (e.g., Adderall, Ritalin, etc.); caffeine (e.g., coffee, cola, etc.); ephedrine (e.g., diet pills, energy drinks, etc.); and eugeroics (e.g., Modafinil, Provigil, etc.) from at least 9:00 AM on Visits 2 and 3
5. Are under treatment for a major injury (e.g., amputation, burns, eye injury, skeletal injury, severe infection, etc.)
6. Have a major medical illness (e.g., active malignancy, cardiovascular disease, diabetes mellitus, HIV, etc.)
7. Are at risk for self-harm determined by a licensed independent practitioner
8. Have indications of recreational substance use determined by a urine drug test
9. Have an abnormal lab value that may indicate major medical illness, which was not cleared by a licensed independent practitioner
10. Have an abnormal lab value that may indicate endocrine dysfunction, which was not cleared by a licensed independent practitioner
11. Have adrenal insufficiency determined by the ACTH stimulation test
12. Have a current bipolar disorder determined by the SCID-IV-TR
13. Have a current psychotic disorder determined by the SCID-IV-TR
14. Have current alcohol dependence determined by the SCID-IV-TR
15. Have current drug dependence determined by the SCID-IV-TR

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10-06; Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-08 (Actual)

PRIMARY OUTCOMES:
Change in NREM time following tesamorelin administration compared to placebo | 1-3 weeks

SECONDARY OUTCOMES:
Within and between group differences in plasma concentration levels of neuroendocrine proteins following tesamorelin administration compared to placebo | 1-3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Gill, Ph.D., Principal Investigator — National Institute of Nursing Research (NINR)